CLINICAL TRIAL: NCT00308425
Title: Effect of Enteric-Coated Mycophenolate Sodium (EC-MPS) Plus Valsartan as Part of Intensified Multi-factorial Intervention Compared to EC-MPS Plus Standard Practice of Care on Development of Transplant Nephropathy in Cadaver Donor Kidney Recipients Given Basiliximab, Cyclosporine Microemulsion (CsA-ME) and Short-term Steroids: a 12-month, Prospective, Randomized, Open-label Multicentre Study (MYTHOS)
Brief Title: Safety and Efficacy of Enteric-coated Mycophenolate Sodium (EC-MPS) Plus Valsartan in Patients With Kidney Transplants (MYTHOS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CERL080A2405IT02
Record Dates: First submitted 2006-03-27; First posted 2006-03-29 (Estimated); Last update posted 2011-01-31 (Estimated); Status verified 2011-01

CONDITIONS: De Novo Renal Transplantation
Keywords: Renal transplantation, EC-MPS
MeSH Terms: interventions — Valsartan

INTERVENTIONS:
Drug: Enteric-coated Mycophenolate sodium (EC-MPS), valsartan

SUMMARY:
The primary aim of this study is to evaluate the safety and efficacy of EC-MPS plus valsartan as part of an intensified multifactorial intervention on the reduction of the 12-month rate of transplant nephropathy compared with EC-MPS plus standard practice of care in recipients of a first cadaver donor kidney transplant given CsA-ME, basiliximab, and short-term steroids.

ELIGIBILITY:
Inclusion criteria

1. Male and female patients aged 18 to 70 years 2. Patients receiving a first kidney transplant from a cadaver donor, who are scheduled to receive CsA-ME and anti-CD25 antibody as primary immunosuppression; 3. Patients able to receive the first dose of EC-MPS within 48 hours of graft reperfusion Exclusion criteria

1. Multi-organ recipients (e.g. kidney and pancreas, double kidney) or previous transplant with any other organ.
2. Recipient of a kidney from a non-heart beating, from a cadaver donor aged more than 70 years, or with cold ischemia time of more than 36 hours
3. Recipient who is HLA-identical to the donor
4. Patients with a PRA level (past or current level) higher than 50%
5. Patients with a known hypersensitivity to EC-MPS or other components of the formulation (e.g. lactose).
6. Patients with thrombocytopenia (< 75,000/mm3), with an absolute neutrophil count of < 1,500/mm3, and/or leukocytopenia (< 2,500/mm3), and/or hemoglobin < 6 g/dL at Screening or Baseline.
7. HIV-positive
8. Positive HBsAg test for both donor and recipients.
9. Unstable angina, acute myocardial infarction or stroke during the last 6 month or heart failure NYHA class III-IV or hemodinamically significant valvular heart disease
10. Liver injury as indicated by transaminase serum levels (ALT and/or AST) greater than 2 x ULN
11. Creatinine kinase (CK) levels greater than 5 x ULN. Additional protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2002-10; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
12-month rate of success in preventing relapse of nephropathy, defined as persistent albumin excretion rate (AER) > 300 mg/24h and safety, compared between groups.

SECONDARY OUTCOMES:
Renal function, as measured by serum creatinine and calculated creatinine clearance after 6 and 12 months;
Glomerular filtration rate (GFR), as plasma clearance of unlabeled iohexol, after 6 and 12 months;
Albumin excretion rate and fractional clearance of albumin after 6 and 12 months;
Fasting blood glucose levels, total cholesterol, triglyceride and HDL levels and systolic and diastolic blood pressure after 6 and 12 months;
Incidence of acute rejection after 6 and 12 months;
Patient and graft survival at 12 months;

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis

REFERENCES:
- [Derived] Natale P, Mooi PK, Palmer SC, Cross NB, Cooper TE, Webster AC, Masson P, Craig JC, Strippoli GF. Antihypertensive treatment for kidney transplant recipients. Cochrane Database Syst Rev. 2024 Jul 31;7(7):CD003598. doi: 10.1002/14651858.CD003598.pub3. PMID 39082471